CLINICAL TRIAL: NCT04418726
Title: The Clinical Value of Intensive Monitoring and Preemptive Intervention in the Maintenance of AVF: a Random Controlled Trial
Brief Title: Intensive Monitoring and Preemptive Intervention in the Maintenance of AVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Bo Shen, Attending Physician, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AVF-assessment
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Vascular Access Malfunction; Vascular Access Complication; Vascular Access Site Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Monitoring and Preemptive Intervention (Experimental): In this group patients receive intensive monitoring and preemptive intervention. AVF surveillance refers to using non-invasive devices to check for the haemodynamic consequences of stenosis by measuring Qa every month. Clinical assessment refers to monitoring for any presence of stenosis by (i) physical examination, by means of visual inspection and presence of abnormal thrill, bruit or pulse and (ii) checking for signs of access dysfunction during dialysis: difficult cannulation, increase in dynamic arterial or venous pressure, inability to achieve the prescribed dialysis blood pump flow (Qb), prolonged bleeding after needle removal, access recirculation or a drop in Kt/V. Preemptive intervention is performed as long as problems are recognized, including health education and timely surgery.
  Interventions: Other: Intensified Monitoring
- Traditional Monitoring and Intervention (No Intervention): In this group patient receive traditional AVF monitoring, includes clinical assessment for any presence of stenosis by (i) physical examination, by means of visual inspection and presence of abnormal thrill, bruit or pulse and (ii) checking for signs of access dysfunction during dialysis: difficult cannulation, increase in dynamic arterial or venous pressure, inability to achieve the prescribed dialysis blood pump flow (Qb), prolonged bleeding after needle removal, access recirculation or a drop in Kt/V.

INTERVENTIONS:
Other: Intensified Monitoring — Apart from clinical assessment, use non-invasive devices to check for the haemodynamic consequences of stenosis by measuring Qa, using either indicator dilution techniques or duplex ultrasound every month.
  Arms: Intensive Monitoring and Preemptive Intervention

SUMMARY:
Whether intensive monitoring and preemptive intervention has an positive clinical effect on arterio-venous fistula (AVF) maintenance is a new issue in hemodialysis (HD) patient management. This study aims to explore the clinical value of intensive monitoring and preemptive intervention on AVF, so to decide the best follow-up items and frequency.

ELIGIBILITY:
Inclusion Criteria:

* patients on HD with AVF in Zhongshan Hospital, Fudan University

Exclusion Criteria:

* with malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
AVF patency rate | 6 months
  AVF patency rate

SECONDARY OUTCOMES:
AVF complication | 12 months
  AVF complication

IPD SHARING:
Plan to Share IPD: No